CLINICAL TRIAL: NCT05595382
Title: Motivations for Stem Cell Transplant Registry Participation
Brief Title: Motivations to Transplant Registry Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Lauren C. Daniel, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro2022000536
Record Dates: First submitted 2022-09-15; First posted 2022-10-27 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: stem cell transplant; bone marrow donor; motivations; altruism
MeSH Terms: conditions — Altruism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Group (Experimental): Participants will be randomly assigned to receive an emotional or rational appeal, stratified by sex.
  Interventions: Behavioral: Emotional Appeal
- Rational Group (Experimental): Participants will be randomly assigned to receive an emotional or rational appeal, stratified by sex.
  Interventions: Behavioral: Rational Appeal

INTERVENTIONS:
Behavioral: Emotional Appeal — Participants will be presented with a short vignette about a child undergoing cancer treatment and needing a bone marrow transplant in order to survive cancer.
  Arms: Emotional Group
Behavioral: Rational Appeal — Participants will be presented with data regarding the importance of considering race/ethnicity when looking for a bone marrow transplant donor and the likelihood of finding a match based on the patient's racial/ethnic background.
  Arms: Rational Group

SUMMARY:
The current study seeks to understand factors that influence college students' likelihood of participating the National Marrow Donor Program (NMDP)/Be the Match for bone marrow and stem cell donations. The secondary aim is to compare emotional and rational approaches to encouraging participation in the registry and how these approaches may impact intentions to participate in the NMDP.

DETAILED DESCRIPTION:
This study is a randomized controlled trial that will randomize participants to receive either an emotional appeal about a child with cancer who needs a bone marrow transplant or a rational appeal using data on the racial/ethnic disparities within the transplant registry.

Participants will be recruited through the Psychology Subject Pool, which will then link students to the study measures in an online survey. Participants will be asked their age to confirm eligibility to participate (students must be between 18-35), and eligible students will be presented with the consent form through the online survey system. Participants will then be asked to complete measures of demographic information, personality/psychological characteristics, and transplant-related knowledge, intentions, and attitudes. All participants will then be given background information on bone marrow transplants.

Randomization: Students will be randomized by sex in the online survey system to the emotional presentation condition or the rational presentation condition. The emotional condition will tell the story of a fictional pediatric patient with cancer who needs a transplant. The rational condition will describe the facts about the need for diversity in the registry.

After being presented with the rational or emotional appeal, participants will again be asked about their intentions to register, their motivations for registering, and their mood.

ELIGIBILITY:
Inclusion Criteria:

* Rutgers Camden Students enrolled in Psych 101 and Method and Theory
* Between the ages of 18-35

Exclusion Criteria:

* Students under 18 years of age or over 36 or older will be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 397 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C Daniel, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University Camden, Camden, New Jersey, United States

REFERENCES:
- [Background] Billen A, Madrigal JA, Scior K, Shaw BE, Strydom A. Donation of peripheral blood stem cells to unrelated strangers: A thematic analysis. PLoS One. 2017 Oct 25;12(10):e0186438. doi: 10.1371/journal.pone.0186438. eCollection 2017. PMID 29069088
- [Background] Butterworth VA, Simmons RG, Bartsch G, Randall B, Schimmel M, Stroncek DF. Psychosocial effects of unrelated bone marrow donation: experiences of the National Marrow Donor Program. Blood. 1993 Apr 1;81(7):1947-59. PMID 8461479
- [Background] CROWNE DP, MARLOWE D. A new scale of social desirability independent of psychopathology. J Consult Psychol. 1960 Aug;24:349-54. doi: 10.1037/h0047358. No abstract available. PMID 13813058
- [Background] Fingrut W, Parmar S, Cuperfain A, Rikhraj K, Charman E, Ptak E, Kahlon M, Graham A, Luong S, Wang YG, Yu J, Arora N, Suppiah R, Li EW, Lee A, Welsh C, Benzaquen M, Thatcher A, Baharmand I, Ladd A, Petraszko T, Allan D, Messner H. The Stem Cell Club: a model for unrelated stem cell donor recruitment. Transfusion. 2017 Dec;57(12):2928-2936. doi: 10.1111/trf.14327. Epub 2017 Sep 24. PMID 28944484
- [Background] Gardner, Paul. (1987). Measuring ambivalence to science. Journal of Research in Science Teaching. 24. 241 - 247. 10.1002/tea.3660240305.
- [Background] Kaster EC, Rogers CR, Jeon KC, Rosen B. Getting to the Heart of Being the Match: A Qualitative Analysis of Bone Marrow Donor Recruitment and Retention Among College Students. Health Educ (Muncie). 2014 Spring;46(1):14-19. PMID 25632376
- [Background] Monaghan M, Yi QL, Green M, Campbell T, Weiss JT, Dibdin N, Mercer D, Elmoazzen H, Allan DS. Factors associated with registrant availability for unrelated adult donor hematopoietic stem cell donation: Analysis of the stem cell registry at Canadian Blood Services. Transfusion. 2021 Jan;61(1):24-28. doi: 10.1111/trf.16129. Epub 2020 Oct 21. PMID 33084098
- [Background] Narayanan P, Wolanskyj A, Ehlers SL, Litzow MR, Patnaik MS, Hogan WJ, Hashmi SK. Medical Students' Knowledge, Familiarity, and Attitudes towards Hematopoietic Stem Cell Donation: Stem Cell Donation Behaviors. Biol Blood Marrow Transplant. 2016 Sep;22(9):1710-1716. doi: 10.1016/j.bbmt.2016.06.014. Epub 2016 Jun 22. PMID 27343721
- [Background] National Marrow Donor Program (2013). Key Figures and Facts. www.bethematch.com
- [Background] Onitilo AA, Lin YH, Okonofua EC, Afrin LB, Ariail J, Tilley BC. Race, education, and knowledge of bone marrow registry: indicators of willingness to donate bone marrow among African Americans and Caucasians. Transplant Proc. 2004 Dec;36(10):3212-9. doi: 10.1016/j.transproceed.2004.10.019. PMID 15686731
- [Background] Rose A, Peters N, Shea JA, Armstrong K. Development and testing of the health care system distrust scale. J Gen Intern Med. 2004 Jan;19(1):57-63. doi: 10.1111/j.1525-1497.2004.21146.x. PMID 14748861
- [Background] Rosenberg, M. (1965). Rosenberg self-esteem scale. Journal of Religion and Health.
- [Background] Rushton, J. P., Chrisjohn, R. D., & Fekken, G. C. (1981). The altruistic personality and the self-report altruism scale. Personality and individual differences, 2(4), 293-302.
- [Background] Surana, P. K., & Lomas, T. (2014). The power of charity: Does giving away money improve the wellbeing of the donor. Indian Journal of Positive Psychology, 5(3), 223-230.
- [Background] Studts JL, Ruberg JL, McGuffin SA, Roetzer LM. Decisions to register for the National Marrow Donor Program: rational vs emotional appeals. Bone Marrow Transplant. 2010 Mar;45(3):422-8. doi: 10.1038/bmt.2009.174. Epub 2009 Aug 3. PMID 19648972
- [Background] Vasconcellos A, Nunes A, Feller E. Knowledge, attitudes, and behaviors regarding the bone marrow registry among college and medical students in Rhode Island. Med Health R I. 2011 Oct;94(10):302-5. No abstract available. PMID 22164662
- [Background] Vekaria KM, Hammell AE, Vincent L, Smith M, Rogers T, Switzer GE, Marsh AA. The role of prospection in altruistic bone marrow donation decisions. Health Psychol. 2020 Apr;39(4):316-324. doi: 10.1037/hea0000819. Epub 2019 Nov 14. PMID 31724423
- [Derived] Daniel LC, Elias G, Shah P, Kokolis N. Increasing participation in the national marrow donor program: A randomized trial. J Health Psychol. 2025 Sep 28:13591053251367869. doi: 10.1177/13591053251367869. Online ahead of print. PMID 41015944

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized after completing study baseline measures. 36 participants dropped out before reaching randomization.
Period: Overall Study
Arm/Group | Emotional Group | Rational Group
Started | 181 | 180
Completed | 181 | 180
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emotional Group | Rational Group | Total
Number analyzed (Participants) | 181 | 180 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.62 (2.62) | 19.71 (2.58) | 19.67 (2.60)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 130 | 131 | 261
  Male | 50 | 49 | 99
  Prefer not to say | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 31 | 26 | 57
  Race/Ethnicity: Black or African American | 28 | 42 | 70
  Race/Ethnicity: Hispanic/Latinx | 32 | 25 | 57
  Race/Ethnicity: Indigenous/Native American | 3 | 0 | 3
  Race/Ethnicity: Middle Eastern | 0 | 3 | 3
  Race/Ethnicity: Native Hawaiian | 0 | 1 | 1
  Race/Ethnicity: White | 52 | 49 | 101
  Race/Ethnicity: More than 1 Race/Ethnicity | 34 | 32 | 66
  Race/Ethnicity: Not reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 181 | 180 | 361

OUTCOME MEASURES:

1. Primary Outcome: Intention to Register
Description: Participants rated the likelihood of registering on a 1-7 scale with higher scores indicating greater intention to join the registry (better outcome). Participants were asked these questions before (baseline) and after (post-intervention) the experimental manipulation.
Time Frame: Baseline and after the experimental manipulation (Post-Intervention)
Population: Likelihood to join registry for all randomized study participants on a 1-7 scale with higher scores indicating a greater likelihood of joining (better outcome).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Emotional Group | Rational Group
Number analyzed (Participants) | 181 | 180
score on a scale
  Baseline | 3.32 (.10) | 3.06 (.104)
  Post-Intervention | 4.15 (0.113) | 3.27 (0.113)
Statistical Analysis 1: Comparison: Emotional Group vs Rational Group; Test type: Superiority — Repeated measures of likelihood to enroll (on a 1 to 7 scale with higher numbers indicating a greater likelihood) pre/post intervention; p = .001, ANOVA; Degrees of freedom (1, 359)

2. Secondary Outcome: Mood
Description: Participant mood was assessed on a 1-10 scale, with higher scores indicating a better mood. Participants were asked these questions before (baseline) and after (post-intervention) the experimental manipulation.
Time Frame: Baseline and after experimental manipulation (Post-Intervention)
Population: Pre/Post Intervention Mood report for randomized participants. 1 did not complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Emotional Group | Rational Group
Number analyzed (Participants) | 181 | 179
units on a scale
  Baseline | 6.59 (.129) | 6.36 (.130)
  Post-Intervention | 6.28 (.137) | 6.18 (.138)
Statistical Analysis 1: Comparison: Emotional Group vs Rational Group; Repeated measures ANOVA comparing mood (rated on a 1-10 scale with higher scores indicating better mood) given to participants before and after the study manipulation by group; Test type: Superiority; p = .357, ANOVA; Degrees of freedom (1, 358)

3. Secondary Outcome: Psychosocial and Demographic Correlates of Intentions to Register--Knowledge
Description: Participants completed a knowledge measure about bone marrow and stem cell transplant donation using true/false statements about transplant donation that was examined as a correlate of their intentions to register with the transplant registry. The measure was scored as a percent of items answered correctly, higher scores indicating better knowledge.
Time Frame: Baseline
Population: Participant knowledge at baseline (pre-intervention) in all randomized participants
Measure: Mean (Standard Deviation); unit: percentage of knowledge items correct
Arm/Group | Emotional Group | Rational Group
Number analyzed (Participants) | 181 | 180
percentage of knowledge items correct | 19.5 (18.0) | 22.6 (18.0)
Statistical Analysis 1: Comparison: Emotional Group vs Rational Group; Test type: Superiority; p = .102, ANOVA

ADVERSE EVENTS:
Time Frame: During the 1 hour study period
Description: Participants could contact the PI with concerns due to study participation.
Arm/Group | Emotional Group | Rational Group
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/181 | 0/180
Other Adverse Events (participants affected / at risk) | 0/181 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05595382/Prot_SAP_000.pdf